CLINICAL TRIAL: NCT00633607
Title: Hereditary Colorectal and Associated Tumor Registry Study
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Randall Brand, Principal Investigator, University of Pittsburgh
Other Study IDs: 04-112
Record Dates: First submitted 2008-03-03; First posted 2008-03-12 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Lynch Syndrome; FAP; Hereditary Diffuse Gastric Cancer; Juvenile Polyposis Syndrome; Peutz-Jeghers Syndrome
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Stomach Neoplasms; Juvenile polyposis syndrome; Peutz-Jeghers Syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Serum, plasma, and extracted DNA are stored for potential future studies.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Research Registry — Information regarding medical and family history is stored in the registry to be used for potential future studies

SUMMARY:
After informed consent, participants will be asked to complete a medical/family history questionnaire and provide a blood sample. Participants will also be asked for their permission for study investigators to access medical records and/or recontact them for updates to their medical and family histories. Data and biospecimens will be stored for potential future research projects.

ELIGIBILITY:
Inclusion Criteria:

* Identified gene mutation
* Personal history of colorectal cancer diagnosed ≤ 50
* Personal history of cancer with tumor studies suggestive of Lynch syndrome
* Personal history of multiple primary tumors associated with a hereditary cancer syndrome (colorectal, uterus, stomach, ovary, small bowel, hepatobiliary tract, transitional cell carcinoma of the renal pelvis/ureter, brain)
* Personal history of one of the above cancers and a family history of one or more of the above cancers
* Personal or family history of diffuse gastric cancer
* From a known genetic predisposition family
* Personal history of > 10 colon adenomas (cumulative over a lifetime)
* Personal history of any number of hamartomatous polyps
* Personal history of multiple large (> 1cm) serrated polyps to right of sigmoid

Exclusion critera:

* Individuals under the age of 8
* Individuals who cannot travel to Pittsburgh for in-person enrollment
* Individuals who cannot provide informed consent

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential research subjects are recruited from our Hereditary GI clinic.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2012-04; Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Establish a Hereditary Colorectal Tumor Registry to facilitate development and implementation of epidemiological, clinical and cancer control research. | 1-N/A (up to 8 years)

CONTACTS AND LOCATIONS:
Overall Officials: Randall E Brand, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States